CLINICAL TRIAL: NCT02506712
Title: Evaluation of Physiological and Biomechanical Efficiency of the PAPAW
Acronym: SmartDrive
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre d'Investigation Clinique et Technologique 805 (Other)
Collaborators: Fondation Garches (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2015-A00758-41
Record Dates: First submitted 2015-07-21; First posted 2015-07-23 (Estimated); Last update posted 2020-09-04 (Actual); Status verified 2017-01

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- spinal cord injury (Experimental): use a wheelchair with and without a assisting device to power manuel wheelchair
  Interventions: Device: SmartDrive assisting device; Device: Standard manuel wheelchair
- volunteer (Other): push a wheelchair with and without a assisting device to power manuel wheelchair
  Interventions: Device: SmartDrive assisting device; Device: Standard manuel wheelchair

INTERVENTIONS:
Device: SmartDrive assisting device — oxygen consumption
Device: Standard manuel wheelchair — oxygen consumption

SUMMARY:
The main objective is to quantify energy expenditure when using the SmartDrive system during manual wheelchair propulsion in external conditions (slope, straight line). For this two comparisons are performed:

Comparison of energy expenditure with and without the use of a system SmartDrive 6 minute propulsion test.

Comparison the risk of musculoskeletal disorders of the wrist during a 6 minute propulsion test.

DETAILED DESCRIPTION:
Prospective study mono-centric, controlled, randomized cross over. Randomization of the equipment (without and with SmartDrive).

22 SCI manual wheelchair users. 22 caregivers (healthy subjects)

ELIGIBILITY:
Inclusion Criteria:

* men and women aged between 18 and 70 years
* spinal cord injury
* having given free and informed consent

Exclusion Criteria:

* No affiliation to a social security scheme
* Refusal to participate in the clinical trial
* Patient under guardianship
* Major cognitive disorder
* Bedsores
* Acute complication or systemic organ

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2015-07-15 (Actual); Primary Completion 2015-10-01 (Actual); Study Completion 2017-10-01 (Actual)

PRIMARY OUTCOMES:
measure of oxygen consumption per unit time (VO2) during propulsion | 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Hugeron, PH, Principal Investigator — Raymond Poincaré Hospital
Locations (1):
- hopital R Poincare, Garches, France